CLINICAL TRIAL: NCT02304744
Title: Utrecht Coronary Biobank (UCORBIO)
Acronym: UCORBIO
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, Crystel Gijsberts, MD, UMC Utrecht
Other Study IDs: 11/183
Record Dates: First submitted 2014-11-26; First posted 2014-12-02 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood and EDTA plasma.
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Observational study, no intervention. — Observational study, no intervention.

SUMMARY:
UCORBIO enrolls patients who undergo coronary angiography (for any indication). The investigators draw blood at the moment of insertion of the procedural arterial catheter.

At the moment of inclusion indication, procedural details, risk factor status, medication use and quality of life (RAND-36 and EuroQoL) is assessed. Patients are then followed-up for the occurrence of major adverse cardiovascular events for 5 years. During the follow-up period patients receive a questionnaire every year to check for hospital admissions. The questionnaires at two and five years of follow-up are enriched with quality of life questionnaires (RAND-36 and EuroQoL).

ELIGIBILITY:
Inclusion Criteria:

* Coronary angiography

Exclusion Criteria:

* Age < 18 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult (>18 years) patients who undergo coronary angiography.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2011-10; Primary Completion 2014-12 (Actual); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
major adverse cardiovascular events [MACE] (Stroke, myocardial infarction, coronary revascularization, death) | 5 years
  Stroke, myocardial infarction, coronary revascularization, death.

CONTACTS AND LOCATIONS:
Locations (1):
- UMC Utrecht, Utrecht, Utrecht, Netherlands

REFERENCES:
- [Derived] Gijsberts CM, Santema BT, Asselbergs FW, de Kleijn DP, Voskuil M, Agostoni P, Cramer MJ, Vaartjes I, Hoefer IE, Pasterkamp G, den Ruijter HM. Women Undergoing Coronary Angiography for Myocardial Infarction or Who Present With Multivessel Disease Have a Poorer Prognosis Than Men. Angiology. 2016 Jul;67(6):571-81. doi: 10.1177/0003319715604762. Epub 2015 Sep 7. PMID 26351289
- [Derived] Gijsberts CM, Agostoni P, Hoefer IE, Asselbergs FW, Pasterkamp G, Nathoe H, Appelman YE, de Kleijn DP, den Ruijter HM. Gender differences in health-related quality of life in patients undergoing coronary angiography. Open Heart. 2015 Aug 27;2(1):e000231. doi: 10.1136/openhrt-2014-000231. eCollection 2015. PMID 26339493
- [Derived] Gijsberts CM, Gohar A, Ellenbroek GH, Hoefer IE, de Kleijn DP, Asselbergs FW, Nathoe HM, Agostoni P, Rittersma SZ, Pasterkamp G, Appelman Y, den Ruijter HM. Severity of stable coronary artery disease and its biomarkers differ between men and women undergoing angiography. Atherosclerosis. 2015 Jul;241(1):234-40. doi: 10.1016/j.atherosclerosis.2015.02.002. Epub 2015 Feb 4. PMID 25670231